CLINICAL TRIAL: NCT04843566
Title: Evaluation of Transperineal Biopsy Under Local Anesthesia, a Novel Approach to Decrease Post-Biopsy Infections and Improve Cancer Detection
Brief Title: PReclude Infection EVEnts With No Prophylaxis Transperineal Biopsy
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20-04021956; 1R01CA241758 (NIH); 18-02-365-NIH (Other: Biomedical Research Alliance of New York (BRANY))
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Infection
Keywords: prostate cancer; prostate biopsy; biopsy infection; fusion biopsy; MRI-targeted biopsy; transperineal; transrectal
MeSH Terms: conditions — Infections; Prostatic Neoplasms | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Men enrolled in this prospective, randomized trial will be randomized in a 1:1 ratio to receive either transperineal MRI-targeted or transrectal MRI-targeted prostate biopsy.
Who Masked: Outcomes Assessor
Masking Description: Radiologists assessing MRI results are blinded to treatment assignment. Pathologists assessing biopsy results are blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transrectal (Active Comparator): Patients will receive a transrectal MRI-guided prostate biopsy.
  Interventions: Procedure: Transrectal MRI-guided prostate biopsy; Drug: Antibiotic (prophylaxis)
- Transperineal (Active Comparator): Patients will receive a transperineal MRI-guided prostate biopsy.
  Interventions: Procedure: Transperineal MRI-guided prostate biopsy

INTERVENTIONS:
Procedure: Transperineal MRI-guided prostate biopsy — Transperineal prostate biopsy will be performed under local anesthesia in the office. This approach avoids transrectal needle tracking.
  Arms: Transperineal
Procedure: Transrectal MRI-guided prostate biopsy — Transrectal prostate biopsy is currently the most popular approach to evaluate a positive screening test for prostate cancer.
  Arms: Transrectal
Drug: Antibiotic (prophylaxis) — For men undergoing transrectal biopsy, antibiotic prophylaxis will be administered in accordance with guidelines from the American Urological Association (AUA).
  No antibiotic prophylaxis will be administered for men undergoing transperineal biopsy.
  Arms: Transrectal

SUMMARY:
Approximately one million transrectal prostate biopsies are performed annually in the U.S., and the risk of post- biopsy infection is increasing due to greater antibiotic resistance of rectal flora. Preliminary data demonstrates that a transperineal MRI-targeted biopsy approach under local anesthesia compared to the standard practice transrectal MRI-targeted prostate biopsy has a much lower risk of infection, comparable pain/discomfort and may improve detection of prostate cancer.

This randomized controlled trial will be the first prospective study to evaluate in-office transperineal MRI targeted prostate biopsy.

The investigators hypothesize that a transperineal MRI-targeted biopsy approach under local anesthesia compared to the standard practice transrectal MRI-targeted prostate biopsy has a much lower risk of infection, comparable pain/discomfort and may improve detection of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the most commonly diagnosed malignancy in U.S. men. There are approximately 1 million prostate biopsy performed annually in the U.S. Almost all biopsies are performed as an office based procedure in under 15 minutes. The precision of biopsy has improved over the last decade with the introduction of MRI guidance/targeting of suspicious lesions within the prostate.

However, significant limitations remain with this approach, including a significantly increasing risk of post-biopsy infection. This arises because more than 97% of all prostate biopsy are performed via a transrectal approach that introduces rectal bacteria with each pass of the biopsy needle into the sterile urinary tract. The current risk of post-transrectal biopsy infection, even with antimicrobial prophylaxis, is high at approximately 7% overall with 3% (30,000 men) requiring hospitalization annually.

Transperineal biopsy is an alternate approach that eliminates the direct introduction of bacteria from the rectum to the prostate. This approach, which is performed without antimicrobial prophylaxis, instead passes the biopsy needle through the perineal skin and pelvic floor.

Transperineal biopsy has not been widely adopted for several reasons. Historically, it has been considered too painful for patients in the clinic and thus was traditionally performed under general anesthesia. The added time, inconvenience and cost has limited its national adoptance. Second, when transrectal biopsy was initially adopted over 40 years ago, antibiotic resistance of rectal flora was not a challenge.

Beyond the potential for in-office transperineal biopsy to significantly reduce or eliminate biopsy infections, transperineal biopsy may also improve cancer detection: studies of transperineal biopsy (performed under general anesthesia) demonstrate higher detection rates for prostate cancer, particularly for anterior zone tumors, compared to transrectal biopsy. This is notable, as anterior tumors are difficult to sample with transrectal. Anterior tumors are also twice as likely to occur in African American men. In fact, our research demonstrates that some of the outcomes disparities in African American men may stem from an underdiagnosis of anterior prostate cancers.

Although transrectal biopsy is used widely, it is associated with a significant and increasing risk of biopsy infections due to growing antibiotic resistance, highlighting the urgent need for a safer alternative approach to prostate biopsy. The study investigators have refined a transperineal approach under local anesthesia with MRI-targeting/guidance without the need for antibiotic prophylaxis. The investigators hypothesize that transperineal MRI targeted biopsy will: (1) largely eliminate post-biopsy infections and costly hospitalizations for urosepsis; (2) be performed in the office with similar discomfort and non-infectious complications compared to transrectal MRI targeted biopsy; and (3) have significantly better detection of prostate cancer.

This multi-center randomized controlled trial will be conducted to evaluate in-office transperineal MRI targeted vs. transrectal MRI targeted biopsy, the current gold standard. This has transformative impact to change current standard of practice.

ELIGIBILITY:
Inclusion Criteria

* Male sex
* Age ≥18 years
* Men without previous prostate biopsy (first time prostate biopsy)
* Willingness to sign informed consent and adhere to the study protocol

Exclusion Criteria

* Acute prostatitis within the last 6 months
* PSA > 20 ng/mL in men who have previously undergone prostate biopsy
* Current non-urologic bacterial infection requiring active treatment with antibiotics
* Unfit to undergo prostate biopsy under local anesthesia
* Prior definitive therapy for prostate cancer, such as radiation therapy or partial gland ablation
* Men who have previously undergone prostate biopsy in whom artifact would reduce quality of prostate MRI (extensive orthopedic pelvic metal)
* Contraindication to prostate MRI (claustrophobia, pacemaker, chronic kidney disease) in men who have previously undergone prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Hu, MD MPH, Principal Investigator — Weill Cornell Medicine, NewYork-Presbyterian
Locations (10):
- United States (10):
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Medical School, Ann Arbor, Michigan
  - NewYork Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - NewYork-Presbyterian Queens, Flushing, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Driscoll CB, Handa N, Huang MM, Murphy AB, Hu JC, Schaeffer EM. Evaluating PI-RADS lesions and clinically significant prostate cancer in Black and Asian men: a PREVENT randomized clinical trial secondary analysis. Prostate Cancer Prostatic Dis. 2025 Nov 26. doi: 10.1038/s41391-025-01057-5. Online ahead of print. PMID 41298852
- [Derived] Driscoll C, Handa N, Huang M, Murphy A, Hu J, Schaeffer E. Evaluating PI-RADS lesions and clinically significant prostate cancer in Black and Asian men: a PREVENT randomized clinical trial secondary analysis. Res Sq [Preprint]. 2025 Jul 4:rs.3.rs-6905600. doi: 10.21203/rs.3.rs-6905600/v1. PMID 40630527

RESULTS

PARTICIPANT FLOW:
Groups:
- Transrectal: Patients will receive a transrectal MRI-guided prostate biopsy.
  Transrectal MRI-guided prostate biopsy: Transrectal prostate biopsy is currently the most popular approach to evaluate a positive screening test for prostate cancer.
  Antibiotic (prophylaxis): For men undergoing transrectal biopsy, antibiotic prophylaxis will be administered in accordance with guidelines from the American Urological Association (AUA).
  No antibiotic prophylaxis will be administered for men undergoing transperineal biopsy.
Period: Overall Study
Arm/Group | Transrectal | Transperineal
Started | 342 | 345
Intent To Treat (Underwent Non-assigned Intervention) | 17 | 12
Completed | 259 | 282
Not Completed | 83 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transrectal | Transperineal | Total
Number analyzed (Participants) | 342 | 345 | 687
Age, Customized [Mean (Full Range); unit: years] | 66 [61 to 71] | 66 [61 to 71] | 66 [61 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 342 | 345 | 687
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 12 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 32 | 76
  White | 168 | 189 | 357
  More than one race | 15 | 17 | 32
  Unknown or Not Reported | 99 | 95 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic: Hispanic ethnicity | 10 | 11 | 21
  Hispanic: Unknown | 332 | 334 | 666
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 342 | 345 | 687

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Experienced Infection, Urinary Retention or Bleeding Requiring Intervention Within 7 Days of Biopsy Based on Transrectal Ultrasound Guided Prostate Biopsy Questionnaire (TRUS-BxQ)
Description: Outcome measure Description Now says: Transrectal Ultrasound Guided Prostate Biopsy Questionnaire (TRUS-BxQ) is a validated biopsy questionnaire that measures adverse events that have occurred due to infection. Patient questionnaires that reported infection complications and duration of symptoms, had their electronic medical records verified to confirm if an infection occurred or not.
Time Frame: 7 days post-biopsy
Population: Subjects in the transrectal arm that underwent a transperineal biopsy or withdrew were excluded from analysis. Subjects in the transperineal arm that underwent a transrectal biopsy or withdrew were excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Transrectal | Transperineal
Number analyzed (Participants) | 280 | 287
percentage of participants
  Infection | 1.4 | 0
  Urinary Retention | 1.1 | 0.3
  Bleeding requiring intervention | 0.4 | 0
Statistical Analysis 1: Comparison: Transrectal vs Transperineal; Infection; Test type: Superiority; p = 0.04, Fisher Exact
Statistical Analysis 2: Comparison: Transrectal vs Transperineal; Urinary retention; Test type: Superiority; p = 0.30, Fisher Exact
Statistical Analysis 3: Comparison: Transrectal vs Transperineal; Bleeding requiring intervention; Test type: Superiority; p = 0.31, Fisher Exact

2. Secondary Outcome: Percentage of Patient Reporting Biopsy Pain and Discomfort
Description: Patient reported pain via a yes/no questionnaire
Time Frame: Immediately following biopsy, 7 days post-biopsy
Population: Subjects in the transrectal arm that underwent a transperineal biopsy or withdrew were excluded from analysis. Subjects in the transperineal arm that underwent a transrectal biopsy or withdrew were excluded from analysis. Any subject that didn't complete a questionnaire was excluded from analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Transrectal | Transperineal
Number analyzed (Participants) | 277 | 283
percentage of participants
  Immediately following biopsy - pain | 3.0 | 3.7
  Immediately following biopsy - discomfort | 3.8 | 4.2
  7-day post biopsy - pain: number analyzed (Participants) | 222 | 226
  7-day post biopsy - pain | 3.6 | 4.5
  7-day post biopsy - discomfort: number analyzed (Participants) | 222 | 226
  7-day post biopsy - discomfort | 1.7 | 2.0
Statistical Analysis 1: Comparison: Transrectal vs Transperineal; Immediately following biopsy - Pain; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Transrectal vs Transperineal; Immediately following biopsy - Discomfort; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Transrectal vs Transperineal; 7-day post biopsy - Pain; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Transrectal vs Transperineal; 7-day post biopsy - Discomfort; Test type: Superiority; p = 0.07, t-test, 2 sided

3. Secondary Outcome: Change in Patient-reported Anxiety, as Measured on a 0-10 Likert Scale
Description: Anxiety will be scored on a 0-10 Likert scale. 0 indicates no anxiety and high scores indicate greater anxiety.
Time Frame: Immediately following biopsy
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transrectal | Transperineal
Number analyzed (Participants) | 279 | 286
score on a scale | 4.2 (2.9) | 3.9 (3.0)
Statistical Analysis 1: Comparison: Transrectal vs Transperineal; Test type: Superiority; p = 0.23, t-test, 2 sided

4. Secondary Outcome: Detection of Clinically Significant Disease as Measured by Gleason Grade Group ≥ 2
Description: Gleason Grade Group is a prostate cancer grading system released by the International Society of Urological Pathology (ISUP). Grade Group 1 indicates Low/Very Low Risk, Grade Group 2 indicates Intermediate (Favorable) Risk, Grade Group 3 indicates Intermediate (Unfavorable) Risk, and Grade Groups 4 and 5 indicate High/Very High Risk.
  Prostate cancer grade will be categorized into insignificant (Gleason Grade Group 1) and clinically significant (Grade Group ≥ 2).
Time Frame: 7 days post-biopsy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Transrectal | Transperineal
Number analyzed (Participants) | 280 | 287
Participants
  Gleason grade group ≥ 2 | 141 | 151
  Gleason grade group 1 | 62 | 49
  No Gleason Score | 77 | 87
Statistical Analysis 1: Comparison: Transrectal vs Transperineal; Gleason grade >=2; Test type: Superiority; p = 0.59, Chi-squared

5. Secondary Outcome: Change in Adverse Events, as Measured on Transrectal Ultrasound Guided Prostate Biopsy Questionnaire (TRUS-BxQ)
Description: Transrectal Ultrasound Guided prostate Biopsy Questionnaire (TRUS-BxQ) is a validated biopsy questionnaire that measures adverse events that have occurred, such as hospital re-admissions, aborted procedures due to discomfort, hematuria, urinary retention, hematospermia, and/or hematochezia. Patient questionnaire consists of Yes/No questions about general complications and duration of adverse events.
Time Frame: 7 days post-biopsy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Transrectal | Transperineal
Number analyzed (Participants) | 280 | 287
Participants
  Infection | 4 | 0
  Urinary Retention | 3 | 1
  Bleeding requiring intervention | 1 | 0
Statistical Analysis 1: Comparison: Transrectal vs Transperineal; Infection; Test type: Superiority; p = 0.04, Fisher Exact
Statistical Analysis 2: Comparison: Transrectal vs Transperineal; Urinary retention; Test type: Superiority; p = 0.30, Fisher Exact
Statistical Analysis 3: Comparison: Transrectal vs Transperineal; Bleeding requiring intervention; Test type: Superiority; p = 0.31, Fisher Exact

ADVERSE EVENTS:
Time Frame: 10 days post biopsy procedure date
Description: Only subjects that were included in the intent to treat analysis were evaluated for adverse events.
Arm/Group | Transrectal | Transperineal
All-Cause Mortality (participants affected / at risk) | 0/280 | 0/287
Serious Adverse Events (participants affected / at risk) | 0/280 | 0/287
Other Adverse Events (participants affected / at risk) | 8/280 | 1/287
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transrectal (N=280) | Transperineal (N=287)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1)
Infection (Renal and urinary disorders) | 4 (4) | 0 (0)
Bleeding (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04843566/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04843566/ICF_000.pdf